CLINICAL TRIAL: NCT03782558
Title: Validation of the Polish Version of the Boston Carpal Tunnel Syndrome Questionnaire
Status: Completed | Type: Observational
Sponsor: Jakub Antczak (Other)
Collaborators: Centrum Neurologii Klinicznej Krakowska Akademia Neurologii (Unknown)
Responsible Party: Sponsor-Investigator, Jakub Antczak, Principal Investigator, Jagiellonian University
Organization: Jagiellonian University (Other)
Other Study IDs: JagiellonianU60
Record Dates: First submitted 2018-12-08; First posted 2018-12-20 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Carpal Tunnel Syndrome
Keywords: carpal tunnel syndrome; pBCTQ; validation; nerve conduction study
MeSH Terms: conditions — Carpal Tunnel Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with CTS: Surgical transection of transverse ligament
  Interventions: Procedure: Surgical transection of transverse ligament

INTERVENTIONS:
Procedure: Surgical transection of transverse ligament — Standard therapy for CTS. An incision is made at the base of the palm of the hand. Then the transverse ligament is cut, which releases the compression of the median nerve and improves the symptoms.
  Other Names: Surgical transection of flexor retinaculum

SUMMARY:
Carpal tunnel syndrome is the most common compression neuropathy. The compression of the median nerve occurs in the carpal tunnel and results in pain and other unpleasant sensations in hand and wrist. In more advanced stage, weakness and wasting of the thenar and other muscles innervated by median nerve occurs, which may lead to permanent impairment of manual performance. The Boston carpal tunnel questionnaire (BCTQ) is one of the most commonly used tools for monitoring of the disease progression and of the effect of therapy. Originally created in English, it has been translated into many languages and subsequently validated. Recently the Polish version has been created and the purpose of this study is to validate it.

DETAILED DESCRIPTION:
Carpal tunnel syndrome (CTS) is the most common compression neuropathy. The compression of the median nerve occurs in the carpal tunnel and results in pain and other unpleasant sensations in hand and wrist. In more advanced stage, weakness and wasting of the thenar and other muscles innervated by median nerve occurs, which may lead to permanent impairment of manual performance. The Boston carpal tunnel questionnaire (BCTQ) (Levine et al. 1993) is one of the most commonly used tools for monitoring of the disease progression and of the effect of therapy. It is a self administered questionnaire, which consists of two subscales, the Symptom severity scale and the Functional status scale. In the first one, the severity of particular symptoms is rated between none or never to very severe or continuous where appropriate. In the second one, the difficulties in performing several typical daily tasks, requiring manual activity is rated between "no difficulty" to "cannot perform activity at all due to hands and wrists symptoms". Originally created in English, it has been translated into many languages and subsequently validated. Recently the Polish version has been created (Polish version of the Boston Carpal Tunnel Questionnaire - pBCTQ) and the purpose of this study is to validate it. The translation from English to Polish has been independently made by two health professionals, native Polish speakers with good acquired knowledge of English. Next, both Polish versions were independently backward-translated to English, by two native English speakers with good acquired knowledge of Polish. Finally, all translators met together and all translations were presented to everyone of them. Possible mistakes in translations from original version into Polish, which might led to discrepancies between backwardly translated versions (from Polish to English) and the original version were discussed and the final version was created. The first step of the study on validation of the Polish version will be the pre-testing. In this step, pBCTQ will be administered to small sample of patients (ten in this study) and the investigators will interview in detail how these participants understand each question of the questionnaire. If pre-testing reveals that patients may understand any question differently from its meaning in the original version, final adjustments will be discussed among the translators and possibly introduced.

The final pBCTQ will be administered before and after surgical treatment to the convenience group of 120 patients with electrodiagnostically confirmed CTS. Moreover, 30 randomly selected patients will be asked to fill out pBCTQ additionally, two weeks after first administration but before surgical treatment. Data from this subgroup will serve to assess the test-retest reliability. pBCTQ will be tested also regarding its consistency, validity and reactivity.

ELIGIBILITY:
Inclusion Criteria:

* Presence of at least one symptom within hand and / or wrist, from the following: paresthesias, sensory loss, tingling, burning sensation, impression of swelling.
* Electrophysiologic confirmation of CTS, which will base on the abnormal latency difference in sensory or motor conduction between median and ulnar nerve or on sensory conduction slowing in median nerve, or on the prolongation of distal motor latency of the median nerve.

(bilateral CTS will be included. pBCTQ will be filled out separately for each hand and the outcomes wil be measured separately for each hand).

Exclusion Criteria:

* Clinical signs or symptoms and /or electrophysiologic results indicative of more generalized peripheral neuropathy.
* Presence of conditions, which may lead to the development of peripheral neuropathy such as diabetes, renal insufficiency, hypothyroidism or amyloidosis.
* Presence of conditions, which may clinically resemble CTS, such as cervical radiculopathy or myelopathy or thoracic outlet syndrome

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited from the patients referred to Krakowska Akademia Neurologii Centrum Neurologii Klinicznej for electrohysiologic verification of their initial, clinical diagnosis of CTS. After the electrophysiology confirms the CTS, the patient will be asked if she/he would like to take part in the study.
Sampling Method: Non-Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2019-01-22 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-09-09 (Actual)

PRIMARY OUTCOMES:
Internal Consistency | Through study completion, an average of six months.
  Consistency between two subscales of pBCTQ (Symptom severity scale and Functional status scale) will be evaluated using Cronbach alfa test.
Validity | Through study completion, an average of six months.
  Validity will be tested by calculating the correlation of the subscore of each of two parts of the questionnaire with the electrophysiologic, six-grade severity level according to Padua et al. (1997).
Reactivity: Correlation between changes in pBCTQ and electrophysiologic severity of CTS | Before treatment and then three months after surgical treatment of CTS
  The reactivity will be evaluated as correlation between change in electrophysiologic severity level of CTS and changes in both pBCTQ subscales after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Jakub Antczak, MD, Principal Investigator — Jagiellonian University
Locations (2):
- Poland (2):
  - Krakowska Akademia Neurologii Centrum Neurologii Klinicznej, Krakow
  - Jagiellonian University Medical College, Krakow

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Padua L, LoMonaco M, Gregori B, Valente EM, Padua R, Tonali P. Neurophysiological classification and sensitivity in 500 carpal tunnel syndrome hands. Acta Neurol Scand. 1997 Oct;96(4):211-7. doi: 10.1111/j.1600-0404.1997.tb00271.x. PMID 9325471
- [Background] Levine DW, Simmons BP, Koris MJ, Daltroy LH, Hohl GG, Fossel AH, Katz JN. A self-administered questionnaire for the assessment of severity of symptoms and functional status in carpal tunnel syndrome. J Bone Joint Surg Am. 1993 Nov;75(11):1585-92. doi: 10.2106/00004623-199311000-00002. PMID 8245050